CLINICAL TRIAL: NCT02224755
Title: Thoratec Corporation MOMENTUM 3, Multi-center Study of MagLev Technology in Patients Undergoing MCS Therapy With HeartMate 3™ IDE Clinical Study Protocol
Brief Title: MOMENTUM 3 IDE Clinical Study Protocol
Acronym: HM3™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC03062014
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Advanced Refractory Left Ventricular Heart Failure
Keywords: Heart Failure; Left Ventricular Assist Device; Ventricular Dysfunction; Cardiomyopathy; Heart Disease; Cardiovascular Disease; Heart-assist devices; Thoratec Corporation
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HeartMate 3 LVAS (HM3 LVAS) (Experimental): Evaluation of the safety and effectiveness of the HeartMate 3 LVAS by demonstrating non-inferiority to the HMII LVAS (HMII) when used for the treatment of advanced, refractory, left ventricular heart failure.
  Interventions: Device: HeartMate 3 LVAS
- HeartMate II LVAS (Active Comparator): Evaluation of the safety and effectiveness of the HeartMate 3 LVAS by demonstrating non-inferiority to the HMII LVAS (HMII) when used for the treatment of advanced, refractory, left ventricular heart failure.
  Interventions: Device: HeartMate II LVAS

INTERVENTIONS:
Device: HeartMate 3 LVAS — Implantation of HeartMate 3 LVAD to evaluate the safety and effectiveness of the HeartMate 3 LVAS by demonstrating non-inferiority to the HMII LVAS (HMII) when used for the treatment of advanced, refractory, left ventricular heart failure
  Arms: HeartMate 3 LVAS (HM3 LVAS)
Device: HeartMate II LVAS — Implantation of the commercially approved HeartMate II LVAD which is the standard treatment for advanced heart failure
  Arms: HeartMate II LVAS

SUMMARY:
The objective of the study is to evaluate the safety and effectiveness of the HM3 LVAS by demonstrating non-inferiority to the HMII LVAS (HMII) when used for the treatment of advanced, refractory, left ventricular heart failure.

DETAILED DESCRIPTION:
The HM3 LVAS is intended to provide hemodynamic support in patients with advanced, refractory left ventricular heart failure; either for short term support, such as a bridge to cardiac transplantation (BTT) or myocardial recovery, or as long term support, such as destination therapy (DT). The HM3 is intended for use inside or outside the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal representative has signed Informed Consent Form (ICF)
2. Age ≥ 18 years
3. BSA ≥ 1.2 m2
4. NYHA Class III with dyspnea upon mild physical activity, or NYHA Class IV
5. LVEF ≤ 25%
6. a) Inotrope dependent OR b) CI < 2.2 L/min/m2, while not on inotropes and subjects must also meet one of the following:

   * On Optimal Medical Management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and are failing to respond
   * Advanced Heart Failure for at least 14 days AND dependent on intra-aortic balloon pump (IABP) for at least 7 days
7. Females of child bearing age must agree to use adequate contraception

Exclusion Criteria:

1. Etiology of heart failure (HF) due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy
2. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator
3. Existence of ongoing mechanical circulatory support (MCS) other than IABP
4. Positive pregnancy test if of childbearing potential
5. Presence of mechanical aortic valve that will not be either converted to a bioprosthesis or oversewn at the time of LVAD implant
6. History of any organ transplant
7. Platelet count < 100,000 x 103/L (< 100,000/ml)
8. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management
9. History of confirmed, untreated AAA > 5 cm in diameter within 6 months of enrollment
10. Presence of an active, uncontrolled infection
11. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy the investigator will require based upon the patients' health status
12. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:

    1. An INR ≥ 2.0 not due to anticoagulation therapy
    2. Total bilirubin > 43 umol/L (2.5 mg/dl), shock liver, or biopsy proven liver cirrhosis
    3. History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, and FEV1 <50% predicted
    4. Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention
    5. History of stroke within 90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 80%) uncorrected carotid stenosis
    6. Serum creatinine ≥ 221 umol/L (2.5 mg/dl) or the need for chronic renal replacement therapy
    7. Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration
13. Patient has moderate to severe aortic insufficiency without plans for correction during pump implant
14. Pre albumin < 150 mg/L (15mg/dL) or Albumin < 30g/L (3 g/dL) (if only one available) ; pre albumin < 150 mg/L (15mg/dL) and Albumin < 30g/L (3 g/dL) (if both available)
15. Planned Bi-VAD support prior to enrollment
16. Patient has known hypo or hyper coagulable states such as disseminated intravascular coagulation and heparin induced thrombocytopenia
17. Participation in any other clinical investigation that is likely to confound study results or affect the study
18. Any condition other than HF that could limit survival to less than 24 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1028 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Crandall, PhD, Study Director — Abbott
Locations (69):
- United States (69):
  - Baptist Health Medical Center - Little Rock, Little Rock, Arkansas
  - Cedars Sinai Medical Center, Beverly Hills, California
  - University of California, San Diego, La Jolla, California
  - Sutter Memorial Hospital, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Hospital @ University of Florida, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health/Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky - Saha Cardiovascular Research Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins Unversity Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Hershey, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas West Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Memorial Hermann Health Systems, Houston, Texas
  - Methodist Houston, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Mehra MR, Naka Y, Uriel N, Goldstein DJ, Cleveland JC Jr, Colombo PC, Walsh MN, Milano CA, Patel CB, Jorde UP, Pagani FD, Aaronson KD, Dean DA, McCants K, Itoh A, Ewald GA, Horstmanshof D, Long JW, Salerno C; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Circulatory Pump for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):440-450. doi: 10.1056/NEJMoa1610426. Epub 2016 Nov 16. PMID 27959709
- [Derived] Sayer G, Ahmed MM, Mehra MR, Gosev I, Vidula H, Devore AD, Horstmanshof DA, Cleveland JC Jr, Stewart GC, Slaughter MS, Mudy K, Wang A, Uriel N. Implantable Cardioverter-Defibrillators and Cardiovascular Resynchronization Therapy with Left Ventricular Assist DevicesA MOMENTUM 3 Trial Analysis. J Card Fail. 2025 Oct;31(10):1548-1557. doi: 10.1016/j.cardfail.2024.12.011. Epub 2025 Jan 22. PMID 39855458
- [Derived] Shah P, Sayer G, Sinha SS, Kanwar MK, Cowger JA, Pagani FD, Nayak A, Mehra MR, Cleveland JC Jr, Psotka MA, Singh R, Desai SS, Lu Q, Hu Y, Connolly A, Kormos RL, Uriel N. Dynamic Risk Estimation of Adverse Events in Ambulatory LVAD Patients: A MOMENTUM 3 Analysis. JACC Heart Fail. 2024 Nov;12(11):1898-1912. doi: 10.1016/j.jchf.2024.05.018. Epub 2024 Jul 24. PMID 39066758
- [Derived] Nayak A, Hall SA, Uriel N, Goldstein DJ, Cleveland JC Jr, Cowger JA, Salerno CT, Naka Y, Horstmanshof D, Crandall D, Wang A, Mehra MR. Predictors of 5-Year Mortality in Patients Managed With a Magnetically Levitated Left Ventricular Assist Device. J Am Coll Cardiol. 2023 Aug 29;82(9):771-781. doi: 10.1016/j.jacc.2023.05.066. PMID 37612008
- [Derived] Mehra MR, Nayak A, Morris AA, Lanfear DE, Nemeh H, Desai S, Bansal A, Guerrero-Miranda C, Hall S, Cleveland JC Jr, Goldstein DJ, Uriel N, Chen L, Bailey S, Anyanwu A, Heatley G, Chuang J, Estep JD. Prediction of Survival After Implantation of a Fully Magnetically Levitated Left Ventricular Assist Device. JACC Heart Fail. 2022 Dec;10(12):948-959. doi: 10.1016/j.jchf.2022.08.002. Epub 2022 Oct 12. PMID 36456068
- [Derived] Uriel N, Milano C, Agarwal R, Lee S, Cleveland J, Goldstein D, Wang A, Crandall D, Mehra MR. Incidence and clinical correlates of de-novo aortic regurgitation with a fully magnetically levitated left ventricular assist device: a MOMENTUM 3 trial portfolio analysis. Eur J Heart Fail. 2023 Feb;25(2):286-294. doi: 10.1002/ejhf.2746. Epub 2022 Nov 29. PMID 36404406
- [Derived] Mehra MR, Goldstein DJ, Cleveland JC, Cowger JA, Hall S, Salerno CT, Naka Y, Horstmanshof D, Chuang J, Wang A, Uriel N. Five-Year Outcomes in Patients With Fully Magnetically Levitated vs Axial-Flow Left Ventricular Assist Devices in the MOMENTUM 3 Randomized Trial. JAMA. 2022 Sep 27;328(12):1233-1242. doi: 10.1001/jama.2022.16197. PMID 36074476
- [Derived] Sheikh FH, Ravichandran AK, Goldstein DJ, Agarwal R, Ransom J, Bansal A, Kim G, Cleveland JC, Uriel N, Sheridan BC, Chomsky D, Patel SR, Dirckx N, Franke A, Mehra MR. Impact of Race on Clinical Outcomes After Implantation With a Fully Magnetically Levitated Left Ventricular Assist Device: An Analysis From the MOMENTUM 3 Trial. Circ Heart Fail. 2021 Oct;14(10):e008360. doi: 10.1161/CIRCHEARTFAILURE.120.008360. Epub 2021 Sep 16. PMID 34525837
- [Derived] Lundgren SW, Florescu DF, Zolty R. Reactivation of Cytomegalovirus Following Left Ventricular Assist Device Implantation: A Case-Control Study. ASAIO J. 2021 Apr 1;67(4):405-410. doi: 10.1097/MAT.0000000000001236. PMID 32740125
- [Derived] Saeed O, Colombo PC, Mehra MR, Uriel N, Goldstein DJ, Cleveland J, Connors JM, Najjar SS, Mokadam NA, Bansal A, Crandall DL, Sood P, Jorde UP. Effect of aspirin dose on hemocompatibility-related outcomes with a magnetically levitated left ventricular assist device: An analysis from the MOMENTUM 3 study. J Heart Lung Transplant. 2020 Jun;39(6):518-525. doi: 10.1016/j.healun.2020.03.001. Epub 2020 Mar 20. PMID 32340871
- [Derived] Patel CB, Blue L, Cagliostro B, Bailey SH, Entwistle JW, John R, Thohan V, Cleveland JC Jr, Goldstein DJ, Uriel N, Su X, Somo SI, Sood P, Mehra MR. Left ventricular assist systems and infection-related outcomes: A comprehensive analysis of the MOMENTUM 3 trial. J Heart Lung Transplant. 2020 Aug;39(8):774-781. doi: 10.1016/j.healun.2020.03.002. Epub 2020 Mar 20. PMID 32276809
- [Derived] Goldstein DJ, Naka Y, Horstmanshof D, Ravichandran AK, Schroder J, Ransom J, Itoh A, Uriel N, Cleveland JC Jr, Raval NY, Cogswell R, Suarez EE, Lowes BD, Kim G, Bonde P, Sheikh FH, Sood P, Farrar DJ, Mehra MR. Association of Clinical Outcomes With Left Ventricular Assist Device Use by Bridge to Transplant or Destination Therapy Intent: The Multicenter Study of MagLev Technology in Patients Undergoing Mechanical Circulatory Support Therapy With HeartMate 3 (MOMENTUM 3) Randomized Clinical Trial. JAMA Cardiol. 2020 Apr 1;5(4):411-419. doi: 10.1001/jamacardio.2019.5323. PMID 31939996
- [Derived] Mehra MR, Uriel N, Naka Y, Cleveland JC Jr, Yuzefpolskaya M, Salerno CT, Walsh MN, Milano CA, Patel CB, Hutchins SW, Ransom J, Ewald GA, Itoh A, Raval NY, Silvestry SC, Cogswell R, John R, Bhimaraj A, Bruckner BA, Lowes BD, Um JY, Jeevanandam V, Sayer G, Mangi AA, Molina EJ, Sheikh F, Aaronson K, Pagani FD, Cotts WG, Tatooles AJ, Babu A, Chomsky D, Katz JN, Tessmann PB, Dean D, Krishnamoorthy A, Chuang J, Topuria I, Sood P, Goldstein DJ; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Left Ventricular Assist Device - Final Report. N Engl J Med. 2019 Apr 25;380(17):1618-1627. doi: 10.1056/NEJMoa1900486. Epub 2019 Mar 17. PMID 30883052
- [Derived] Colombo PC, Mehra MR, Goldstein DJ, Estep JD, Salerno C, Jorde UP, Cowger JA, Cleveland JC Jr, Uriel N, Sayer G, Skipper ER, Downey FX, Ono M, Hooker R Jr, Anyanwu AC, Givertz MM, Mahr C, Topuria I, Somo SI, Crandall DL, Horstmanshof DA. Comprehensive Analysis of Stroke in the Long-Term Cohort of the MOMENTUM 3 Study. Circulation. 2019 Jan 8;139(2):155-168. doi: 10.1161/CIRCULATIONAHA.118.037231. PMID 30586698
- [Derived] Mehra MR, Salerno C, Naka Y, Uriel N, Cleveland JC, Horstmanshof D, Goldstein DJ; MOMENTUM 3 Investigators. A tale of the twist in the outflow graft: An analysis from the MOMENTUM 3 trial. J Heart Lung Transplant. 2018 Nov;37(11):1281-1284. doi: 10.1016/j.healun.2018.08.011. Epub 2018 Aug 24. No abstract available. PMID 30245150
- [Derived] Mehra MR, Salerno C, Cleveland JC, Pinney S, Yuzefpolskaya M, Milano CA, Itoh A, Goldstein DJ, Uriel N, Gulati S, Pagani FD, John R, Adamson R, Bogaev R, Thohan V, Chuang J, Sood P, Goates S, Silvestry SC. Healthcare Resource Use and Cost Implications in the MOMENTUM 3 Long-Term Outcome Study. Circulation. 2018 Oct 30;138(18):1923-1934. doi: 10.1161/CIRCULATIONAHA.118.035722. PMID 29807933
- [Derived] Mehra MR, Goldstein DJ, Uriel N, Cleveland JC Jr, Yuzefpolskaya M, Salerno C, Walsh MN, Milano CA, Patel CB, Ewald GA, Itoh A, Dean D, Krishnamoorthy A, Cotts WG, Tatooles AJ, Jorde UP, Bruckner BA, Estep JD, Jeevanandam V, Sayer G, Horstmanshof D, Long JW, Gulati S, Skipper ER, O'Connell JB, Heatley G, Sood P, Naka Y; MOMENTUM 3 Investigators. Two-Year Outcomes with a Magnetically Levitated Cardiac Pump in Heart Failure. N Engl J Med. 2018 Apr 12;378(15):1386-1395. doi: 10.1056/NEJMoa1800866. Epub 2018 Mar 11. PMID 29526139
- [Derived] Goldstein DJ, Mehra MR, Naka Y, Salerno C, Uriel N, Dean D, Itoh A, Pagani FD, Skipper ER, Bhat G, Raval N, Bruckner BA, Estep JD, Cogswell R, Milano C, Fendelander L, O'Connell JB, Cleveland J; MOMENTUM 3 Investigators. Impact of age, sex, therapeutic intent, race and severity of advanced heart failure on short-term principal outcomes in the MOMENTUM 3 trial. J Heart Lung Transplant. 2018 Jan;37(1):7-14. doi: 10.1016/j.healun.2017.11.001. Epub 2017 Nov 3. PMID 29154131
- [Derived] Cowger JA, Naka Y, Aaronson KD, Horstmanshof D, Gulati S, Rinde-Hoffman D, Pinney S, Adatya S, Farrar DJ, Jorde UP; MOMENTUM 3 Investigators. Quality of life and functional capacity outcomes in the MOMENTUM 3 trial at 6 months: A call for new metrics for left ventricular assist device patients. J Heart Lung Transplant. 2018 Jan;37(1):15-24. doi: 10.1016/j.healun.2017.10.019. Epub 2017 Oct 24. PMID 29153637
- [Derived] Uriel N, Colombo PC, Cleveland JC, Long JW, Salerno C, Goldstein DJ, Patel CB, Ewald GA, Tatooles AJ, Silvestry SC, John R, Caldeira C, Jeevanandam V, Boyle AJ, Sundareswaran KS, Sood P, Mehra MR. Hemocompatibility-Related Outcomes in the MOMENTUM 3 Trial at 6 Months: A Randomized Controlled Study of a Fully Magnetically Levitated Pump in Advanced Heart Failure. Circulation. 2017 May 23;135(21):2003-2012. doi: 10.1161/CIRCULATIONAHA.117.028303. Epub 2017 Apr 6. PMID 28385948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 69 study sites in the United States from 2014 to 2016.
Groups:
- HeartMate II (Intent-to-Treat): Patients randomized to HeartMate II LVAS (control device)
- HeartMate 3 (Intent-to-Treat): Patients randomized to HeartMate 3 LVAS
Period: Randomization to Device Implant
Arm/Group | HeartMate II (Intent-to-Treat) | HeartMate 3 (Intent-to-Treat)
Started | 512 (Patients in the Full Study Cohort (n=1028) who were randomized to HeartMate II) | 516 (Patients in the Full Study Cohort (n=1028) who were randomized to HeartMate 3)
Completed | 505 (Patients who underwent HeartMate II LVAS implant) | 515 (Patients who underwent HeartMate 3 LVAS implant)
Not Completed | 7 | 1
Not completed — Withdrawn prior to implant | 7 | 1
Period: Two Year Follow up Post-implant
Arm/Group | HeartMate II (Intent-to-Treat) | HeartMate 3 (Intent-to-Treat)
Started | 505 | 515
Completed | 247 | 289
Not Completed | 258 | 226
Not completed — Death | 103 | 98
Not completed — Heart transplant | 137 | 119
Not completed — Device explant or permanent deactivation | 3 | 3
Not completed — Withdrawn post-implant | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HeartMate II (Intent-to-Treat) | HeartMate 3 (Intent-to-Treat) | Total
Number analyzed (Participants) | 512 | 516 | 1028
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 59 (12) | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 105 | 198
  Male | 419 | 411 | 830
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or ethnic group: White | 367 | 342 | 709
  Race or ethnic group: Black | 120 | 145 | 265
  Race or ethnic group: Asian | 3 | 8 | 11
  Race or ethnic group: Native Hawaiian or Pacific Islander | 4 | 0 | 4
  Race or ethnic group: Other | 18 | 21 | 39
Ischemic Cause of Heart Failure [Count of Participants; unit: Participants] | 240 | 216 | 456
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 238 | 215 | 453
History of Stroke [Count of Participants; unit: Participants] | 56 | 50 | 106
Intended Goal of Support [Count of Participants; unit: Participants]
  Bridge to transplantation | 121 | 113 | 234
  Bridge to candidacy for transplantation | 81 | 86 | 167
  Destination therapy | 310 | 317 | 627
Inotropes [Count of Participants; unit: Participants] | 423 | 445 | 868
Implantable cardioverter-defibrillator [Count of Participants; unit: Participants] | 382 | 352 | 734
Intra-aortic balloon pump [Count of Participants; unit: Participants] | 79 | 64 | 143
INTERMACS profile [Count of Participants; unit: Participants] — INTERMACS profiles describe the clinical profile of advanced heart failure patients who may be candidates for mechanical circulatory support. There are 7 profiles ranging from Profile 1 (most sick) to Profile 7 (least sick). Profile 1 indicates critical cardiogenic shock. Profile 2 indicates progressive decline. Profile 3 indicates stable but inotrope dependent. Profile 4 indicates resting symptoms. Profile 5 indicates exertion intolerant. Profile 6 indicates exertion limited. Profile 7 indicates advanced NYHA Class 3 (clinically stable with a reasonable level of comfortable activity).
  Participants
    1 | 18 | 11 | 29
    2 | 146 | 156 | 302
    3 | 251 | 272 | 523
    4 | 82 | 67 | 149
    5-7 or not provided | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Short Term Primary End Point
Description: Survival at 6 months free of disabling stroke (Modified Rankin Score > 3) or reoperation to replace or remove a malfunctioning device
Time Frame: The first 294 randomized Subjects will be followed for 6 months or to outcome (transplant, explant, or death), whichever occurs first.
Population: First 294 randomized Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate II (Intent-to-Treat) | HeartMate 3 (Intent-to-Treat)
Number analyzed (Participants) | 142 | 152
Participants | 109 | 131
Statistical Analysis 1: Comparison: HeartMate II (Intent-to-Treat) vs HeartMate 3 (Intent-to-Treat); Test type: Non-Inferiority — Non-inferiority would be demonstrated if the 95% lower confidence boundary for the difference between treatment groups (HM3 - HMII) in the occurrence of the primary end point would be greater than -10 percentage points, at a one-sided alpha level of 0.025 or a two-tailed P value of less than 0.05; p < 0.001, Farrington-Manning risk difference; Risk Difference (RD) = 9.4, 95% CI 1-sided [lower limit -2.1]

2. Primary Outcome: Long Term Primary End Point
Description: Survival at 2 years free of disabling stroke (Modified Rankin Score > 3) or reoperation to replace or remove a malfunctioning device
Time Frame: The first 366 randomized Subjects will be followed for 24 months or to outcome (transplant, explant, or death), whichever occurs first.
Population: First 366 randomized Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate II (Intent-to-Treat) | HeartMate 3 (Intent-to-Treat)
Number analyzed (Participants) | 176 | 190
Participants | 106 | 151
Statistical Analysis 1: Comparison: HeartMate II (Intent-to-Treat) vs HeartMate 3 (Intent-to-Treat); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Farrington-Manning risk difference; Risk Difference (RD) = 19.2, 95% CI 1-sided [lower limit 9.8]

3. Secondary Outcome: Powered Secondary End Point: Pump Replacement at Two Years
Description: In addition to powering the study on the primary endpoints for PMA approval, the study will pre-specify a powered secondary endpoint to evaluate incidence of pump replacements at 24 months. HeartMate II is the control.
Time Frame: As they occur up to 24 months or to Outcome, whichever occurs first
Population: All subjects who underwent implant with the assigned device
Measure: Count of Participants; unit: Participants
Groups:
- HeartMate II (As-Treated): Subjects randomized to HeartMate II LVAS who underwent implant with the assigned device
- HeartMate 3 (As-Treated): Subjects randomized to HeartMate 3 LVAS who underwent implant with the assigned device
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
Participants | 57 | 12
Statistical Analysis 1: Comparison: HeartMate II (As-Treated) vs HeartMate 3 (As-Treated); Based on data in the Sponsor's device tracking database, 7% of patients with the HeartMate II LVAS receive a pump replacement by 24 months. The expected proportion of patients with the HeartMate 3 LVAS to receive a pump replacement by 24 months was assumed to be 3%. We estimated that to demonstrate superiority of HeartMate 3 to HeartMate II with a power of 80% and α = 0.05 (2-sided), a total of 1028 patients (514 per arm) were required using the Fisher's exact test; Test type: Superiority; p < 0.001, Fisher Exact; Risk Ratio (RR) = 0.21, 95% CI 2-sided [.11 to .38]

4. Secondary Outcome: EuroQoL 5D-5L (EQ-5D-5L) Total Score
Description: Quality of Life as measured by EuroQoL 5 Dimension-5 Level (EQ-5D-5L) total score. The EQ-5D-5L questionnaire has patients rate their quality of life across 5 categories of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scores from the 5 dimensions are summed for the total score which ranges from 5 to 25 with higher scores indicating more problems and a worse quality of life.
Time Frame: Baseline to 24 months
Population: Analysis population only includes patients still ongoing on LVAD support at the specified time periods who completed the assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
score on a scale
  Baseline: number analyzed (Participants) | 475 | 486
  Baseline | 11.2 (4.4) | 11.1 (4.3)
  6 months: number analyzed (Participants) | 385 | 418
  6 months | 8.5 (3.2) | 8.5 (3.3)
  24 months: number analyzed (Participants) | 227 | 275
  24 months | 9.2 (3.8) | 8.8 (3.6)

5. Secondary Outcome: EuroQol-5D-5L Visual Analogue Scale
Description: Quality of life as measured by the visual analogue scale from the EuroQol-5D-5L questionnaire. The patient rates their current state of health with the visual analogue scale. The scale ranges from 0 to 100. Higher scores indicate a better quality of life.
Time Frame: Baseline to 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
score on a scale
  Baselline: number analyzed (Participants) | 475 | 486
  Baselline | 48 (25) | 50 (24)
  6 months: number analyzed (Participants) | 386 | 420
  6 months | 74 (19) | 76 (18)
  24 months: number analyzed (Participants) | 227 | 276
  24 months | 75 (19) | 76 (19)

6. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). Scores range from 0 to 100. Higher scores indicate better quality of life and fewer heart failure symptoms.
Time Frame: Baseline to 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
score on a scale
  Baseline: number analyzed (Participants) | 482 | 493
  Baseline | 40 (23) | 39 (20)
  6 months: number analyzed (Participants) | 388 | 421
  6 months | 70 (21) | 70 (20)
  24 months: number analyzed (Participants) | 227 | 277
  24 months | 68 (23) | 69 (22)

7. Secondary Outcome: Six Minute Walk Test
Description: Functional status as measured by the Six Minute Walk Test. The Six Minute Walk Test measures the distance a patient is able to walk during 6 minutes without running or jogging.
Time Frame: Baseline to 24 months
Population: Analysis population only includes patients still ongoing on LVAD support at the specified time periods who completed the assessment. Patients unable to walk due to heart failure symptoms were assigned a distance of zero.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
meters
  Baseline: number analyzed (Participants) | 452 | 471
  Baseline | 129 (156) | 136 (160)
  6 months: number analyzed (Participants) | 333 | 365
  6 months | 327 (136) | 310 (142)
  24 months: number analyzed (Participants) | 174 | 211
  24 months | 361 (337) | 323 (156)

8. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: Functional status as measured by NYHA classification. NYHA class categorizes patients by the severity of their heart failure symptoms. As the class increases, the degree of symptoms is more severe indicating worse functional status. Class I indicates no limitation of physical activity. Class II indicates slight limitation of physical activity. Class IIIA indicates marked limitation of physical activity where less than ordinary physical activity causes fatigue, palpitation, dyspnea, or angina pain. Class IIIB indicates marked limitation of physical activity where mild physical activity causes fatigue, palpitation, dyspnea, or angina pain. Class IV indicates inability to carry on any physical activity without discomfort.
Time Frame: Baseline to 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
Participants
  Class I or II at Baseline: number analyzed (Participants) | 504 | 514
  Class I or II at Baseline | 0 | 0
  Class I or II at 6 Months: number analyzed (Participants) | 392 | 428
  Class I or II at 6 Months | 310 | 340
  Class I or II at 24 Months: number analyzed (Participants) | 229 | 275
  Class I or II at 24 Months | 176 | 219

9. Secondary Outcome: Rehospitalizations
Description: Rate of all cause rehospitalization
Time Frame: From initial discharge to two years post-implant
Population: Analysis population only includes Subjects who were discharged on LVAD support from the implant hospitalization
Measure: Number; unit: events per patient year
Groups:
- HeartMate II (As-Treated): Subjects randomized to HeartMate II LVAS who underwent implant with the assigned device and were discharged on LVAD support
- HeartMate 3 (As-Treated): Subjects randomized to HeartMate 3 LVAS who underwent implant with the assigned device and were discharged on LVAD support
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 471 | 485
events per patient year | 2.47 | 2.26

10. Secondary Outcome: Adverse Event Rates
Description: Events-per-patient-year (EPPY) for anticipated adverse events as defined in the study protocol
Time Frame: Two years post-implant
Measure: Number; unit: events per patient year
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
Number analyzed (Participants) | 505 | 515
events per patient year
  Arterial Non-CNS Thromboembolism | 0.02 | 0.01
  Bleeding | 0.95 | 0.61
  Cardiac Arrhythmia | 0.45 | 0.37
  Hepatic Dysfunction | 0.04 | 0.03
  Hypertension | 0.08 | 0.07
  Major Infection | 0.82 | 0.82
  Myocardial Infarction | 0.01 | 0.01
  Stroke | 0.18 | 0.08
  Hemorrhagic Stroke | 0.07 | 0.03
  Ischemic Stroke | 0.11 | 0.04
  Debilitating Stroke | 0.07 | 0.04
  Other Neurological Event | 0.08 | 0.09
  Pericardial Fluid Collection | 0.07 | 0.04
  Psychiatric Episode | 0.07 | 0.08
  Renal Dysfunction | 0.08 | 0.11
  Respiratory Failure | 0.17 | 0.19
  Right Heart Failure | 0.23 | 0.27
  RVAD | 0.03 | 0.03
  Venous Thromboembolism | 0.04 | 0.04
  Wound Dehiscence | 0.02 | 0.01
  Suspected Device Thrombosis | 0.12 | 0.01
  Hemolysis | 0.01 | 0.01

ADVERSE EVENTS:
Time Frame: Two years post-implant
Arm/Group | HeartMate II (As-Treated) | HeartMate 3 (As-Treated)
All-Cause Mortality (participants affected / at risk) | 103/505 | 98/515
Serious Adverse Events (participants affected / at risk) | 466/505 | 483/515
Other Adverse Events (participants affected / at risk) | 235/505 | 261/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HeartMate II (As-Treated) (N=505) | HeartMate 3 (As-Treated) (N=515)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 10 | 5
Bleeding (Blood and lymphatic system disorders) | 271 | 214
Cardiac Arrhythmia (Cardiac disorders) | 174 | 149
Hepatic Dysfunction (Hepatobiliary disorders) | 23 | 20
Hypertension (Vascular disorders) | 18 | 23
Major Infection (Infections and infestations) | 251 | 274
Myocardial Infarction (Cardiac disorders) | 5 | 6
Stroke (Nervous system disorders) | 98 | 51
Other Neurological Event (Nervous system disorders) | 47 | 59
Pericardial Fluid Collection (Cardiac disorders) | 44 | 25
Psychiatric Episode (Psychiatric disorders) | 24 | 31
Renal Dysfunction (Renal and urinary disorders) | 52 | 70
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 94 | 110
Right Heart Failure (Cardiac disorders) | 127 | 151
Venous Thromboembolism (Vascular disorders) | 14 | 20
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 8 | 4
Suspected Device Thrombosis (Product Issues) | 70 | 7
Hemolysis (Blood and lymphatic system disorders) | 8 | 6
Other (General disorders) | 277 | 340
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HeartMate II (As-Treated) (N=505) | HeartMate 3 (As-Treated) (N=515)
Bleeding (Blood and lymphatic system disorders) | 26 | 31
Cardiac Arrhythmia (Cardiac disorders) | 46 | 54
Hypertension (Vascular disorders) | 29 | 19
Major Infection (Infections and infestations) | 79 | 95
Psychiatric Episode (Psychiatric disorders) | 21 | 24
Right Heart Failure (Cardiac disorders) | 19 | 28
Other Adverse Event (General disorders) | 113 | 139

LIMITATIONS AND CAVEATS:
This was a non-blinded study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MOMENTUM 3 has a study specific charter that governs the overall publication and presentation policy for all abstracts and manuscripts related to MOMENTUM 3 clinical data.

DOCUMENTS (2):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02224755/Prot_001.pdf
  • Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT02224755/SAP_000.pdf